CLINICAL TRIAL: NCT04371354
Title: Outcomes After Implementation of a Protective Protocol for Covid-19 in Large Spanish Endoscopy Units.
Brief Title: Outcomes of Covid-19 Protective Measures in Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Principal Investigator, Juan J Vila, MD, PhD, medical doctor, University of Navarra associate professor, Fundacion Miguel Servet
Other Study IDs: 2020-COCHE
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Covid-19 Disease; Endoscopy Unit
Keywords: Covid-19 disease; endoscopy; gastrointestinal; personal protective equipment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study evaluating the outcomes of implementation of a protective protocol for Covid-19 for patients and staff in a large endoscopy unit.

DETAILED DESCRIPTION:
Detailed description: SARS-Covid-19 virus pandemic has had a big impact both socially and on operation of health facilities. During the Covid-19 outbreak most of the scheduled endoscopies were cancelled and only emergent and urgent endoscopies were performed in the unit. This meant that for six weeks, around 98% of our daily workload was cancelled. During that time the investigators have developed a protocol in order to resume scheduled endoscopic activity in the decreasing phase of the pandemic.

The hypothesis of this prospective observational study is that implementation of a protocol based upon Covid PCR tests and clinical triage is useful to categorize two types of Covid-19 infection risk and two levels of personal protection equipments required.

The primary aim is to evaluate the outcomes of implementing a protective protocol with two levels of protection for Covid-19 in the endoscopy unit. As secondary aims, the investigators, want to evaluate the endoscopy unit staff and patients infection rate after implementation of the protective protocol; and the utility of previous Covid PCR testing and on day clinical triage to discriminate patients before endoscopy.

A brief daily questionnaire will be filled by all the endoscopy unit staff members questioning about type of procedures performed in their allocated endoscopy room, level of protection used and PCR status of their attended patients. Patients will be followed up for a period of two weeks to discard development of Covid-19 disease with possible origin in their visit to the endoscopy unit.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing an endoscopic procedure with written informed consent given.
* Staff allocated in the endoscopy unit.

Exclusion Criteria:

* Refection to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing an endoscopic procedure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-12-27 (Estimated)

PRIMARY OUTCOMES:
Rate of new Covid infection of patients and staff members | 3 months
  Number of new Covid infection of patients and staff members

SECONDARY OUTCOMES:
Covid disease prevalence in the patients referred to endoscopy | 3 months
  Number of patients referred to endoscopy with Covid disease
Categorization by clinical triage and Covid Test | 3 months
  Categorization of patients by clinical triage and Covid Test
Type of endoscopy procedure and staff protective equipment | 3 months
  Influence of the type of endoscopy procedure and staff protective equipment

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Vila, PhD, Principal Investigator — Tertiary referral hospital: Complejo Hospitalario de Navarra. Pamplona.Spain
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No